CLINICAL TRIAL: NCT05428319
Title: Expression of STEAP-1 and p40 in Prostatic Carcinoma and Its Mimickers: An Immunohistochemical Study
Brief Title: Expression of STEAP-1 and p40 in Prostatic Carcinoma and Its Mimickers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aliaa Bakr Ahmed, Assistant lecturer, Sohag University
Other Study IDs: Soh-Med-22-06-14
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Prostatic Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prostatic carcinoma is the second most common cancer in men with high incidence of morbidity and mortality. It is a common health problem. Most cases occur at the age of 50 years, reaching its peak at 60-70 years of age. Diagnosis of prostatic carcinoma is still a problematic issue as accurate diagnosis can be very challenging due to the presence of either a small focus of cancer or the presence of many benign mimickers of malignancy.

Six transmembrane epithelial antigen of the prostate 1 (STEAP-1) is primarily localized at the cell membrane, mostly at cell-cell junctions, but it may also be found dispersed in the cytoplasm. In prostate, the expression of STEAP-1 is higher in neoplastic tissues compared to its restricted expression in normal prostatic samples.

The antibody designated as p40 recognizes exclusively ΔNp63 and not TAp63. In prostate tissues, it has been shown that p40, the ΔNp63 isoform of p63, stains prostatic basal cells as reliable as p63 in most cases. Furthermore, aberrant staining of tumor cells was seen more rarely with p40 than with p63.

In this study, the investigators hope to solve some problematic issues in diagnosis of prostatic carcinoma and reach the better way to distinguish prostatic carcinoma from mimicking lesions by using both STEAP-1 and p 40. Also, the way to detect cancer at early stage of development and its progression which is extremely important as it allows establishing the most effective treatment and predicting patient's outcome.

ELIGIBILITY:
Inclusion Criteria:

* Trans-rectal ultrasound guided biopsy (TRUS) procedure, transurethral resection prostatectomy (TURP) and radical prostatectomy.
* Prostatic adenocarcinoma and prostatic lesions that mimic prostatic adenocarcinoma

Exclusion Criteria:

* Patients with recurrence of the primary tumor.
* Patients with a history of preoperative chemotherapy and/or radiotherapy.
* Insufficient or tiny tissue biopsies

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: Formalin-fixed and paraffin embedded prostatic tissue blocks from 70 patients
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Prostatic Carcinoma | One or two days after staining sections with the markers
  Immunohistochemical Expression of STEAP-1 and p40 in Prostatic carcinoma and mimickers

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Bakr, Principal Investigator — Faculty of medicine, Sohag University
Locations (1):
- Aliaa Bakr Ahmed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided